CLINICAL TRIAL: NCT04141111
Title: ADJUST: Impact of Professional Continuous Glucose Monitoring in People With Insulin-treated Type 2 Diabetes
Brief Title: Retrospective and Prospective Study on Professional Continuous Glucose Monitoring in Insulin-treated Type 2 Diabetes
Acronym: ADJUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associacao Protectora dos Diabeticos de Portugal (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 639/2015
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Evaluation of clinical outcomes and patient reported outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CGM intervention (Experimental): Underwent intervention defined by the intermittent use of a continuous glucose monitoring (CGM) device.
  Interventions: Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) — On each visit (baseline, 4, 8, and 12 months), participants received an iPro2 CGM device (MiniMed Medtronic), placed according to the manufacturer's standard procedure. The iPro2 was used each time for 7-days. During this period, patients were asked to perform 4 SMBG measurements daily for calibration (fasting, lunch, dinner, and before bed). Patients received a diary to register food intake, physical activity and medication, SMBG values, and any diabetes-related event (extra consultations, phone calls, etc) in the previous 4 months.
  Each time, CGM data was interpreted by an expert clinician, and a report was delivered, within one week, to the respective healthcare team. This report was discussed together by the patient and one member of the healthcare team, either in consultation or by phone, agreeing on any necessary therapeutic changes. If necessary, extra consultations for nutrition, nursing, or education, were scheduled, to address specific needs identified during rCGM review.

SUMMARY:
In people with type 2 diabetes (T2D) without adequate glycemic control for an extended period of time, continuous glucose monitoring (CGM) can provide detailed information about daily glycemic profile facilitating therapeutic adjustments decision which can contribute to an improvement of glycemic control and overall health status.

The ADJUST study aims to evaluate the impact of CGM systems' use on clinical decision and glycemic control of people with badly controlled T2D, already under insulin therapy.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a growing health problem worldwide. The PrevaDiab study, which studied the prevalence of diabetes in Portugal in 2010, estimated a prevalence of 11.7 %, representing about 905 000 patients with diabetes. Taking the demographic evolution of the Portuguese population, these estimates were updated in 2015, and the global prevalence is expected to have risen to 13.3 % of the adult population.

The International Diabetes Federation (idf) recommends the following glycaemia levels: <100 mg dL-1 (eq 5.6 mmol L-1) for impaired fasting glucose and <140 mg dL-1 (eq 7.8 mmol L-1) for 2h glycaemia. Several guidelines recommend frequent glucose measurements as an integral part of the patients' education and self-monitoring.

The percentage of glycated haemoglobin (HbA1c) is used as a long-term glycaemic control proxy, as it gives the mean value of the previous 3 months blood glycose concentrations. idf recommends a maximum 6.5 % HbA1c concentration for all diabetic patients - 7.0 % for type II diabetes mellitus (dm-ii) patients - and, the closer to this value, the fewer risk of complications. The American Diabetes Association (ADA) recommends at least two HbA1c measures per year in controlled patients and three times per year in patients with therapeutic changes and/ or failures.

According with Sartore and collaborators, glucose variability indicators describe the glucose profile of diabetic patients and identify any worsening glycaemic control more accurately than HbA1c tests. However, the capillary glycaemic measure - the standard monitoring blood glucose (smbg) - has some issues that can compromise the optimal diabetes management: with smbg, blood glucose measures are more intermittent, are insufficient to evaluate the glycaemic profile of the patient, and it does not show what happens between two measurements. This situation makes it difficult to interpret and extrapolate information necessary to make adequate decisions in the therapeutic adjustments.

Another clinical important issue is concerned with hypoglycaemia. Hypoglycaemia events limit the efficacy of intensive insulin therapy, especially in patients with great glucose variability, and are associated with increased risk of diabetic complications and cardiovascular disease. The smbg ideal frequency is difficult to establish and consequently, hypo and hyperglycaemic events may be underestimated, even when the measurements and done more frequently than recommended. This underestimation of glucose fluctuations may constitute a critical problem as they have a potential important role in the long term complications occurrence. Several studies report the efficacy of using a professional continuous glucose monitoring (pCGM) device on the detection and reduction of hypoglycaemia and on the detection of hyperglycaemia, alone or compared with SMBG.

Another important parameter is the area under the curve (AUC) in hypoglycaemia, that is, taking into account not only the duration of the events but also its severity.

This information may be crucial for the provider to make clinical decisions and perform therapeutic adjustment in order to control glucose levels more efficiently. Additionally, with a better control of the disease, fewer events are expected to occur showing not only a better clinical situation but also economic benefits of the pCGM over the SMBG alone.

The iPro2 is a pCGM device (from Medtronic Minimed, Northridge, CA) intended to continuously record interstitial glucose levels in persons with dm. It is also intended to be worn for intermittent periods to uncover glycaemic variability and patterns. The data obtained can then be used to maximize treatment strategies to improve patient outcomes.

The study's primary objective is to compare the difference in mean glycated haemoglobin level after clinical decision on diabetes treatment based on pCGM.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to enrolment.
* Male or female, aged between 18-65 years old.
* Type 2 Diabetes Mellitus for more than 12 months, on insulin, on a stable dose for 60 days prior to screening.
* Available clinical records for the past 12 months, regarding medical treatment for diabetes and A1c evaluations.
* A1c >7.5 % in the 60 days prior to screening.
* Discrepancies between A1c and glycaemic levels (the log book not reflecting the A1c result) that justify the clinical decision of pCGM future use.
* Decision to use Carelink iPro must precede enrollment.
* Ability to adhere to protocol requirements.

Exclusion Criteria:

* Gestational Diabetes.
* Pregnant or planning to become pregnant during the course of the study.
* Continuous Glucose Monitoring use by any device or manufacturer in the year prior to screening.
* Serious or unstable medical or psychological condition which, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Inability to comply with study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-03-22 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Glycemic control | -12 months to 12 months, in relation to study initiation
  Evaluated by glycated haemoglobin (A1c). A1c is expressed as %, in relation to native haemoglobin. This is a validated clinical laboratory parameter.
Glycemic control | Study initiation and 4, 8 and 12 months
  Evaluated by TIR (time-in-range), deduced through CGM-generated analysis as the time spent between 70 and 140 mg/dl glucose. TIR is expressed as % of time duration.

SECONDARY OUTCOMES:
Health status | Study initiation and 12 months
  Evaluated by the Global Health Questionnaire (GHQ-12). Results range between 0 and 36. A GHQ score above 24 indicates psychological distress.
Treatment satisfaction | Study initiation and 12 months
  Evaluated by the Diabetes Treatment Satisfaction Questionnaire (DTSQ). Satisfaction is calculated by the partial sum (questions 1,4,5,6,7,8) designated DTSQS. Results range from 0 to 36. A DTSQS partial score below 23 indicates low treatment satisfaction.
Therapeutic changes | During the previous year, and at 4, 8 and 12 months
  Frequency and characteristics (drug, dosage and duration) of therapeutic regimen adjustments. Drugs are registered by commercial name and active principle. Dosage is registered as mg or international units, as adequate.

CONTACTS AND LOCATIONS:
Overall Officials: Joao Raposo, MD PhD, Study Director — Associacao Protectora dos Diabeticos de Portugal
Locations (1):
- APDP, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ribeiro RT, Andrade R, Nascimento do O D, Lopes AF, Raposo JF. Impact of blinded retrospective continuous glucose monitoring on clinical decision making and glycemic control in persons with type 2 diabetes on insulin therapy. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1267-1275. doi: 10.1016/j.numecd.2020.12.024. Epub 2020 Dec 31. PMID 33612381